CLINICAL TRIAL: NCT04827823
Title: Five-year Retrospective Clinical Evaluation of Multi-surface Amalgam and Resin Composite Restorations Placed by Dental Students
Brief Title: Retrospective Evaluation of Posterior Direct Restorations
Status: Completed | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 109006
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-03

CONDITIONS: Dental Caries Class II
Keywords: Amalgam, Dental; Composite Resin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1- Amalgam restorations: Multi-surface amalgam restorations performed by dental students and are in function for about 5 years.
  Interventions: Other: Retrospective evaluation of amalgam and composite restorations
- Group 2- Composite restorations: Multi-surface composite restorations performed by dental students and are in function for about 5 years.
  Interventions: Other: Retrospective evaluation of amalgam and composite restorations

INTERVENTIONS:
Other: Retrospective evaluation of amalgam and composite restorations — Multi-surface restorations that were performed by dental students and that are in function for the last five years will be clinically evaluated with mirrors and probes according to the modified USPHS criteria.

SUMMARY:
This retrospective study aims to evaluate the clinical performance of posterior multi-surface Class II amalgam (AM) and resin composite (RC) restorations placed by dental students over a five-year period.

DETAILED DESCRIPTION:
Purpose: The aim of this retrospective study is to evaluate the clinical performance of posterior multi-surface Class II amalgam (AM) and resin composite (RC) restorations placed by dental students over a five-year period. Materials and Methods: A total of 119 multi-surface Class II restorations (three or more surfaces) placed by third and fourth year students will be evaluated (AM: n = 69 and RC: n = 50). Restorations were assessed clinically according to the USPHS criteria by two independent evaluators using mirrors and probes. Data will be analyzed using Chisquare, Mann-Whitney and Wilcoxon tests at a 0.05 level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Presence of multi-surface (three or more surfaces) composite or amalgam restorations placed by dental students over a five-year period.

Exclusion Criteria:

* Children
* Restorations performed before or after five years on the time of evaluation
* Restorations with fewer than 3 surfaces

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults patients who had complex amalgam or resin composite restorations (three or more surfaces) placed on molar or premolar areas by dental students in the Adult Dental Clinic over a five-year period.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Postoperative sensitivity | 5 years
  No Patient-reported sensitivity to hot and cold stimuli, sweets, clenching, and chewing related to the restoration (Alpha)
Secondary caries | 5 years
  No visual evidence of dark, deep discoloration adjacent to the restoration (Alpha)
Proximal contact | 5 years
  No open contact. Contact offers resistance to the dental floss (Alpha)
Marginal Adaptation | 5 years
  Restoration closely adapted to the tooth. No crevice visible (Alpha)
Fracture restoration | 5 years
  No evidence of fracture (Alpha)
Fracture tooth | 5 years
  No evidence of fracture (Alpha)
Anatomy | 5 years
  Restorations continuous with existing anatomic form (Alpha)

CONTACTS AND LOCATIONS:
Locations (1):
- Schulich Medicine and Dentistry - Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cetin AR, Unlu N, Cobanoglu N. A five-year clinical evaluation of direct nanofilled and indirect composite resin restorations in posterior teeth. Oper Dent. 2013 Mar-Apr;38(2):E1-11. doi: 10.2341/12-160-C. Epub 2012 Dec 5. PMID 23215545
- [Result] Mjor IA, Jokstad A. Five-year study of Class II restorations in permanent teeth using amalgam, glass polyalkenoate (ionomer) cerment and resin-based composite materials. J Dent. 1993 Dec;21(6):338-43. doi: 10.1016/0300-5712(93)90006-c. PMID 8258583
- [Result] Vidnes-Kopperud S, Tveit AB, Gaarden T, Sandvik L, Espelid I. Factors influencing dentists' choice of amalgam and tooth-colored restorative materials for Class II preparations in younger patients. Acta Odontol Scand. 2009;67(2):74-9. doi: 10.1080/00016350802577800. PMID 19085213
- [Result] Correa MB, Peres MA, Peres KG, Horta BL, Barros AD, Demarco FF. Amalgam or composite resin? Factors influencing the choice of restorative material. J Dent. 2012 Sep;40(9):703-10. doi: 10.1016/j.jdent.2012.04.020. Epub 2012 Apr 28. PMID 22546263
- [Result] Rasines Alcaraz MG, Veitz-Keenan A, Sahrmann P, Schmidlin PR, Davis D, Iheozor-Ejiofor Z. Direct composite resin fillings versus amalgam fillings for permanent or adult posterior teeth. Cochrane Database Syst Rev. 2014 Mar 31;(3):CD005620. doi: 10.1002/14651858.CD005620.pub2. PMID 24683067
- [Result] Rho YJ, Namgung C, Jin BH, Lim BS, Cho BH. Longevity of direct restorations in stress-bearing posterior cavities: a retrospective study. Oper Dent. 2013 Nov-Dec;38(6):572-82. doi: 10.2341/12-432-C. Epub 2013 Apr 3. PMID 23550914
- [Result] Beck F, Lettner S, Graf A, Bitriol B, Dumitrescu N, Bauer P, Moritz A, Schedle A. Survival of direct resin restorations in posterior teeth within a 19-year period (1996-2015): A meta-analysis of prospective studies. Dent Mater. 2015 Aug;31(8):958-85. doi: 10.1016/j.dental.2015.05.004. Epub 2015 Jun 16. PMID 26091581
- [Result] Borgia E, Baron R, Borgia JL. Quality and Survival of Direct Light-Activated Composite Resin Restorations in Posterior Teeth: A 5- to 20-Year Retrospective Longitudinal Study. J Prosthodont. 2019 Jan;28(1):e195-e203. doi: 10.1111/jopr.12630. Epub 2017 May 17. PMID 28513897